CLINICAL TRIAL: NCT00378040
Title: Toronto Vascular Disease Risk Factor Assessment Program: Systematic Assessment of Vascular Risk
Brief Title: Systematic Assessment of Vascular Risk
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Thomas Lindsay, Professor of Surgery, University Health Network, Toronto
Other Study IDs: 01-541S
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is hypothesized that patients with vascular disease are undertreated for modifiable risk factors, leading to increased morbidity and mortality in this population.

The objective of this study is to develop a comprehensive database that will demonstrate the current adequacy of risk factor management in this high risk population, and that will provide needed guidance for future treatment options.

ELIGIBILITY:
Inclusion Criteria:

All patients who attend the Vascular Surgery Clinic at Toronto General Hospital, St. Michael's Hospital, and St. Joseph's Health Centre who have PAD, cerebrovascular disease (CBVD), or aneurysms will be eligible for this study. Patients who are currently enrolled in other clinical studies are eligible for this study; however proper adherence to the other study will take precedence over of the current proposal.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with confirmend PAD
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lindsay, M.D, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
See JAMA Surgery 2016 epublished First Author Dr M Hussain